CLINICAL TRIAL: NCT01590927
Title: Reliability and Validation of 3-D Electromagnetic Tracking During Pelvic Floor Muscle (PFM) Activation - a Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Moser, Helene (Individual)
Responsible Party: Principal Investigator, Helene Moser, Physiotherapist, Moser, Helene
Other Study IDs: MScPTHM
Record Dates: First submitted 2012-04-27; First posted 2012-05-03 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Pelvic Floor Dyssynergia
Keywords: pelvic floor; ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 20 healthy women

SUMMARY:
Now a days the ultrasound is seen as a valid and reliable measurement tool to test the Pelvic Floor Muscle (PFM) movement (Sherburn, Murphy, Carroll, Allen, & Galea, 2005). The hypothesis is that the electromagnetic tracking system, TrakSTARTM, can measure the PFM movement in an equal or even more precise way. The TrakSTARTM will have the advantage to be used in measuring functional movements. In this Master thesis the hypothesis is to show a good reliability by trampoline jumping (physical activity).

DETAILED DESCRIPTION:
There will be two measurements. One measurement of MVIC and quick flicks will be done in a standing and supine position with 3 repetitions. The TrakSTARTM, Ultrasound, surface EMG and Accelerometer will measure the PFM movements and activation simultaneously. The Ultrasound is measured from one tester (to guaranty a high intratester reliability) (Sherburn et al., 2005).

TrakSTARTM, surface EMG and Accelerometer will measure 3 Trampoline jumps. The measurements will be done once during one hour. The women will insert the vaginal probe by themselves and stay dressed during the measurement procedure. The measurements will be done in a standardized way. All the arrangements are made to ensure the hygiene requirements.

ELIGIBILITY:
Inclusion Criteria:

* women
* aged between 18 and 35 years
* anamnestically healthy
* nulliparous and
* a BMI between 18 and 30

Exclusion Criteria:

* latex and nickel allergy
* anamnestically current pregnancy
* menstruation
* urogenital operations
* anal operations
* vaginal infections

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy women, students of the University of Applied Sciences Health
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-02 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
the way in x-y coordinates for the pelvic floor mouvement measured by the ultrasonography and TrakSTAR | one year
  the mouvement of the pelvic floor is measured similtanous by the ultrasound and the TrakSTAR

SECONDARY OUTCOMES:
EMG | one year
  EMG will measure the contraction of the plevic floor

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Radlinger, PhD, Study Chair — Berner Fachhochschule Gesundheit, Bern, Switzerland
Locations (1):
- Inselspital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Peng Q, Jones RC, Constantinou CE. 2D Ultrasound image processing in identifying responses of urogenital structures to pelvic floor muscle activity. Ann Biomed Eng. 2006 Mar;34(3):477-93. doi: 10.1007/s10439-005-9059-3. Epub 2006 Feb 16. PMID 16496082
- [Background] Sherburn M, Murphy CA, Carroll S, Allen TJ, Galea MP. Investigation of transabdominal real-time ultrasound to visualise the muscles of the pelvic floor. Aust J Physiother. 2005;51(3):167-70. doi: 10.1016/s0004-9514(05)70023-4. PMID 16137242